CLINICAL TRIAL: NCT04573153
Title: A Multi Centre, Randomised, Controlled, Open-Label Phase 2/3 Study to Evaluate the Efficacy, Tolerability and Safety of Metabolic Cofactor Supplementation and Hydroxychloroquine Combination in Covid-19 Patients
Brief Title: Metabolic Cofactor Supplementation and Hydroxychloroquine Combination in Covid-19 Patients
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Planned enrollment was not fulfilled.
Sponsor: ScandiBio Therapeutics AB (Industry)
Collaborators: Istanbul Medipol University Hospital (Other); Istanbul Umraniye Training and Research Hospital (Unknown); Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government); Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government); Bagcilar Training and Research Hospital (Other Government); Kanuni Sultan Suleyman Training and Research Hospital (Other); Alanya Alaaddin Keykubat University Alanya Training and Research Hospital (Unknown); Canakkale 18 Mart University Health Research and Application Hospital (Unknown); Monitor CRO (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COVID-19-MCS
Record Dates: First submitted 2020-09-30; First posted 2020-10-05 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2020-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; Sorbitol

STUDY DESIGN:
Intervention Model Description: This study was planned as a parallel group, randomized and open label study. The subjects will be randomized on a 3:1 basis to the cofactor supplementation combination plus hydroxychloroquine treatment or hydroxychloroquine +placebo treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm (Experimental): Subjects in ambulatory-at home-treatment will receive hydroxychloroquine (standard therapy) + dietary supplement consisting of serine, L-carnitine tartrate, N-acetylcysteine and nicotinamide riboside.
  Interventions: Drug: Hydroxychloroquine + Metabolic cofactor supplementation
- Placebo Arm (Placebo Comparator): Subjects will take hydroxychloroquine (standard therapy) + dietary supplement placebo.
  Interventions: Drug: Hydroxychloroquine + Sorbitol

INTERVENTIONS:
Drug: Hydroxychloroquine + Metabolic cofactor supplementation — Treatment arm will include dietary supplement consisting of serine, L-carnitine tartrate, N-acetylcysteine and nicotinamide riboside + standard therapy (hydroxychloroquine).
  Arms: Treatment Arm
Drug: Hydroxychloroquine + Sorbitol — Placebo comparator will include sorbitol as placebo + standard therapy (hydroxychloroquine).
  Arms: Placebo Arm

SUMMARY:
This open label, randomized, controlled, investigator-initiated, multi-centre trial aims to establish metabolic improvements in COVID-19 subjects by dietary supplementation with cofactors N-acetylcysteine, L-carnitine tartrate, nicotinamide riboside and serine plus standard therapy. The primary objective is to assess the clinical efficacy of the combination of metabolic cofactors supplementation and hydroxychloroquine in COVID-19 patients.

DETAILED DESCRIPTION:
Coronaviruses are a large family of ribonucleic acid viruses that cause mild to moderate upper respiratory diseases in humans. There is an urgent need for COVID-19 therapeutics due to the S-shaped curve expansion of the infections, widespread pandemic status, and global burden. Given the similarities between SARS-CoV-2 and other coronaviruses, and its relative ease of sample acquisition and study, it has been widely accepted that drug repositioning is a promising approach to make available an effective, safety-assured treatment in a timely manner.

This open label, randomized, controlled, investigator-initiated, multi-centre trial aims to establish metabolic improvements in COVID-19 subjects by dietary supplementation with cofactors N-acetylcysteine, L-carnitine tartrate, nicotinamide riboside and serine plus standard therapy. The investigational drug products, the mixture of the four co-factors will be administered as a powder with strawberry aroma to be dissolved in 200 ml of preferably cold still drinking water and be consumed within 5 minutes.

This study is planned as a Phase II / III clinical drug research to be conducted in patients diagnosed with COVID-19. Patients will be ambulatory and after the diagnosis/confirmation of diagnosis, will be sent home with their treatment. However, patients may be hospitalised during this initial examination period due to deterioration in their physical health or due to any medical condition which was not present at admission.

The primary objective is to assess the clinical efficacy of the combination of metabolic cofactors supplementation and hydroxychloroquine in COVID-19 patients. For the primary purpose, the proportion of patients who were hospitalised during the course of disease until 14 days after the initial diagnosis of Covid-19 disease will be compared. Patients who were hospitalised during the 14-day period, but at any time point after consenting will be evaluated as an end-point occurrence.

The secondary aim in this study is to evaluate the safety and tolerability of metabolic cofactors supplementation and hydroxychloroquine combination.

The initial part of the Phase II/III study is planned as a Phase II study which will enrol 100 patients and after an interim analysis it will conclude as a Phase III study (300 patients). Totally 400 COVID-19 disease patients will be randomized on a 3:1 basis to the combination metabolic cofactors supplementation and hydroxychloroquine or hydroxychloroquine+ placebo in eight clinical sites in Turkey.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders (females and males) over 18 years of age
* Written informed consent obtained from the subjects prior to any procedures related to the study
* Understand all procedures to be applied within the scope of the study protocol
* Ambulatory patients with symptoms diagnosed with COVID-19 with Chest tomography (CT) result positivity in the last 72 hours
* Patients with stable clinical course and who could be treated on an ambulatory basis.

Exclusion Criteria:

* Patients who has partial oxygen saturation below 93% and require immediate hospitalisation after diagnosis
* Patients, upon initial examination, decided to be hospitalised at the intensive care-unit
* Inability or unwillingness to give written informed consent
* At physicians decision, the trial involvement will not be in patients' best interest, or any condition that does not allow the protocol to be followed safely
* Patients considered as inappropriate for this study for any reason
* Active participation in another clinical study
* Uncontrolled Type 1 or type 2 diabetes
* Severe liver disease (e.g. Child Pugh score ≥ C, AST>5 times upper limit)
* Patients with known severe renal impairment (estimated glomerular filtration rate ≤30 mL/min/1.73 m2) or receiving continuous renal replacement therapy, hemodialysis, peritoneal dialysis
* Significant cardiovascular co-morbidity (i.e. heart failure)
* Patients with phenylketonuria (contraindicated for NAC)
* Known allergy for substances used in the study
* Pregnant or breastfeeding patients, or patients with positive pregnancy test in a pre-dose examination
* Receipt of any experimental treatment for COVID-19 within the 30 days prior to the time of the screening evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
The evaluation of clinical efficacy of the combination of metabolic cofactor supplementation and hydroxychloroquine | 14 days
  The clinical efficacy will be evaluated by comparing the proportion of patients who were hospitalised during the course of disease until 14 days after the initial diagnosis of Covid-19.

SECONDARY OUTCOMES:
Adverse Event (AE), Serious Adverse Event (SAE) and discontinuation of treatment | 14 days
  Number/characteristics of Adverse Event (AE), Serious Adverse Event (SAE) and discontinuation of treatment due to study drug from baseline until the end of study.
Chest Tomography | 1 day
  Chest imaging will be documented at baseline visit.
ECG Measurement | 1 day
  Change in heart rate will be measured at baseline visit.
Change of complete blood count from baseline | 14 days
  Complete blood count includes number of blood cells and concentration of hemoglobin. Complete blood count will be performed to measure possible toxic effects of the metabolic cofactors supplementation and hydroxychloroquine combination on hematological system.
Changes in alanine aminotransferase (ALT) levels from baseline | 14 days
  Clinical evaluation of ALT levels from baseline until the end of study.
Changes in aspartate aminotransferase (AST) levels from baseline | 14 days
  Clinical evaluation of AST levels from baseline until the end of study.
Changes in C-reactive protein (CRP) levels from baseline | 14 days
  Clinical evaluation of CRP levels from baseline until the end of study.
Changes in creatinine levels from baseline | 14 days
  Clinical evaluation of creatinine levels from baseline until the end of study.
Changes in D-dimer levels from baseline | 14 days
  Clinical evaluation of D-dimer levels from baseline until the end of study.
Changes in ferritin levels from baseline | 14 days
  Clinical evaluation of ferritin levels from baseline until the end of study.
Changes in triglycerides levels from baseline | 14 days
  Clinical evaluation of triglycerides levels from baseline until the end of study.
Changes in LDH levels from baseline | 14 days
  Clinical evaluation of LDH levels from baseline until the end of study.

CONTACTS AND LOCATIONS:
Overall Officials: Assoc. Prof. Levent DOĞANAY, MD, Principal Investigator — University of Health Sciences Istanbul Ümraniye Training and Research Hospital
Locations (1):
- University of Health Sciences Istanbul Ümraniye Training and Research Hospital, Istanbul, Turkey (Türkiye)